CLINICAL TRIAL: NCT04185740
Title: The Stability in Medication Responsiveness During Research Experiments in Parkinson's Disease
Brief Title: Medication Responsiveness in Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Alice Nieuwboer, Principal Investigator, KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: S62564
Record Dates: First submitted 2019-11-26; First posted 2019-12-04 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Parkinson Disease; Medication Compliance; Tapping Task; Smartphone
MeSH Terms: conditions — Parkinson Disease; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Home-based validation (Experimental): The home-based validation of the TTT will give insight in the task performance of patients OFF-medication compared to ON-medication and on different time points in the medication cycle during 7 days
  Interventions: Device: CloudUPDRS - Tapping Task

INTERVENTIONS:
Device: CloudUPDRS - Tapping Task — The TTT, consisting of two targets, will be presented on the screen of the smartphone. Participants will be instructed to alternate between the two targets using their index finger for 30 seconds. The task will always be performed with the left hand first and then with the right hand. The touch-sensitive screen of the smartphone will measure the timing of each touch event, its duration, the coordinates on the phone screen and the amount of pressure applied.

SUMMARY:
Up till now, dopaminergic replacement is considered as the gold standard for the symptomatic treatment of motor symptoms in Parkinson's disease (PD). However, the intake, especially higher doses when taken for a longer duration, are associated with several side effects including response fluctuations. These fluctuations in medication response are often characterized by a wearing-OFF period, also defined as the recurrence of PD symptoms before a patient should take the next dose of medication. The duration of test sessions during research experiments (e.g. in the field of rehabilitation) can interfere with the period of the optimal therapeutic effect of dopaminergic medication, influencing outcomes of a study. Therefore, the objective of this project is to get more insight in the measurability of ON-OFF fluctuations by testing the applicability of a short and simple timed tapping task (TTT) on a smartphone in rehabilitation research studies. The assessment can be useful for future clinical studies in PD where a precise estimation of medication is indispensable for accurate research outcomes.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of PD, based on the UK Brain Bank Diagnostic Criteria
* Hoehn & Yahr stage I-III
* Mini Mental State Examination (MMSE) scores >24
* Right-handedness
* No other known disease or disorder that will interfere with the experiments

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-07-25 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2020-10-20 (Actual)

PRIMARY OUTCOMES:
Tap frequency | 7 days
  Taps per second
Mean hand movement time between taps | 7 days
  Inter-tap time in milliseconds
Actual distance between taps | 7 days
  Inter-tap distance in centimeters
Visual analogue scale (VAS) | 7 days
  To indicate the subjective medication responsiveness (current golden standard to measure medication fluctuations)

CONTACTS AND LOCATIONS:
Overall Officials: Alice Nieuwboer, Principal Investigator — KU Leuven
Locations (1):
- Department of Rehabilitation Sciences, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Stamate, C., et al., The cloudUPDRS app: A medical device for the clinical assessment of Parkinson's Disease. Pervasive and Mobile Computing, 2018. 43: p. 146-166.
- [Derived] Broeder S, Roussos G, De Vleeschhauwer J, D'Cruz N, de Xivry JO, Nieuwboer A. A smartphone-based tapping task as a marker of medication response in Parkinson's disease: a proof of concept study. J Neural Transm (Vienna). 2023 Jul;130(7):937-947. doi: 10.1007/s00702-023-02659-w. Epub 2023 Jun 2. PMID 37268772